CLINICAL TRIAL: NCT02051712
Title: Cardiovascular Effects of Preferred Home-based Exercise Training and Extended Adherence Measures in Systolic Heart Failure - Pilot Study
Brief Title: Cardiovascular Effects of Preferred Home-based Exercise Training in Systolic Heart Failure
Acronym: HOMEX-HF-P
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DZHK-HGW-001
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; exercise training; preferred training; prevention
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care (No Intervention): Usual car accruing to guidelines
- Individualized training (Experimental): Individualized exercise training program in addition to usual care
  Interventions: Behavioral: exercise training
- Individualized training plus adherence measures (Experimental): Individualized exercise training plus measures to increase adherence
  Interventions: Behavioral: exercise training; Behavioral: Adherence measures

INTERVENTIONS:
Behavioral: exercise training — individualized exercise training
  Arms: Individualized training; Individualized training plus adherence measures
Behavioral: Adherence measures — Measures to increase adherence to exercise training
  Arms: Individualized training plus adherence measures

SUMMARY:
The aim of the study is I. To assess whether an individualized exercise training program is superior as compared to usual care with respect to exercise tolerance, II. to assess whether intervention tools that aim to increase exercise adherence are superior to an individualized exercise training alone with respect to exercise tolerance and long-term effects, and III. to identify biomarkers that that may be implemented into novel intervention tools aiming to increase exercise adherence in patients with chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* women and men
* age 30-75 years
* chronic heart failure (NYHA II/III), left ventricular ejection fraction ≤40% be echo
* disease duration ≥ 6 month
* medical therapy accruing to guidelines (drug, devices, including CRT)
* written informed consent

Exclusion Criteria:

* acute myocarditis
* instable angina
* heart surgery (e.g. ICD implantation, bypass) with last 6 weeks; CRT implantation within the last 6 months before study start
* severe cardiovascular events (myocardial infarction, cardiac decompensation, ICD shock, PCI due to instable angina) < 6 weeks before study start
* preplanned hospital admission or intervention (e.g. planned revascularization, ICD implantation)
* uncorrected valve regurgitation or stenosis (> second degree)
* safety concerns regarding or other reasons against exercise training
* severe depression
* regular exercise training within the last 6 weeks
* life expectancy < 1 year

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-02; Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
VO2@AT | Month 9
  Change of cardiopulmonary exercise tolerance from baseline to 9 month follow-up measured by exercise testing: oxygen uptake at anaerobic threshold per kg body weight (METs)

SECONDARY OUTCOMES:
Training adherence | 9, 12, 18 and 24 month
  Adherence to training sessions

OTHER OUTCOMES:
AE | 9, 12, 18 and 24 month
  Adverse events, related and unrelated to exercise training

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Dörr, MD, Principal Investigator — University Greifswald
Locations (1):
- Marcus Dörr, Greifswald, Germany